CLINICAL TRIAL: NCT01971775
Title: Clinical Study for Energy Based Devices in Open Gastrectomy for Gastric Cancer: Conventional Monopolar Electrosurgery vs. Ultrasonically Activated Shear(UAS)
Brief Title: Clinical Study for Energy Based Devices in Open Gastrectomy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Johnson & Johnson Medical Companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENERGY_FRM001480
Record Dates: First submitted 2011-09-18; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Cancer
Keywords: Ultrasonically Activated Shear; Conventional Monopolar Electrocautery; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ultrasonically Activated Shear (Active Comparator): Dissection and lymphovascular sealing with Ultrasonically Activated Shears
  Interventions: Device: Ultrasonically activated Shears
- Conventional Monopolar Electrocautery (Active Comparator): Dissection and lymphovascular sealing with Conventional Monopolar Electrocautery
  Interventions: Device: Conventional Monopolar Electrocautery

INTERVENTIONS:
Device: Ultrasonically activated Shears — Dissection and lymphovascular sealing with Ultrasonically Activated Shears
  Other Names: Harmonic Scalpel, Ethicon Endo-Surgery, INC (USA)
  Arms: Ultrasonically Activated Shear
Device: Conventional Monopolar Electrocautery — Dissection and lymphovascular sealing with Conventional Monopolar Electrocautery
  Other Names: Monopolar Electrocautery
  Arms: Conventional Monopolar Electrocautery

SUMMARY:
Surgery is the first standard treatment for stomach cancer, but it still has negative factors such as bleeding, leakage, closure, surgery part infection and cardiovascular and lung complication by general anesthesia.

electric cautery is used extensively in surgery room due to the utility of simultaneous severance and hemostasis. In some case, the electric current from vitality electrode may unexpectedly stimulate or damage nearby muscles and nerves. Ultrasonically activated shears (UAS) is a device to transform the protein of organ for organ incision or hemostasis. General advantages possibly include shortened operating time, decrease of operative blood loss, and relatively less damages to the normal organ. UAS is commonly used in the operation room, which is now considered as a secure and useful medical device for for tissue dissection and coagulation. Also, it is expected to lower the risk of surgery by reducing operating time and blood loss.

However, clinical evidence is not sufficient for this device until now. Therefore, in this study,

1. Evaluate the utility, efficacy, and safety of energy based device, in the case of open gastrectomy
2. Would like to compare the following two kinds of energy based devices. A. For conventional monopolar electrosurgery group : dissection and sealing will be conducted by conventional monopolar electrocautery device B. For UAS group : dissection and sealing will be conducted by UAS

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven primary gastric adenocarcinoma
* Patients who may undergo distal gastrectomy
* Patients who qualified for open gastrectomy for gastric cancer stage T1-3, M0 according to the 7th International Union Against Cancer classification
* 20 ≤ age ≤ 75
* Patients with informed consent

Exclusion Criteria:

1. Previous abdominal operation Hx.
2. Patients who are impossible to undergo Billroth-I reconstruction because of duodenal invasion caused by duodenal ulcers or gastric cancer
3. Patients who have CT defined ascites prior to operation
4. Patients with liver dysfunction defined as T.Bil>1.2 or albumin<3.0
5. Patients with heart disease such as uncontrolled hypertension, history of angina or coronary artery disease, history of cardiomyopathy, Ventricular Ejection Fraction <50% measured by echocardiography
6. Patients with renal dysfunction defined as creatinine>1.4 mg/dL or Blood Urea Nitrogen>26mg/dL
7. Patients with severe pulmonary dysfunction defined as Forced Expiratory Volume at 1 second<1.0 L in Pulmonary Function Test
8. Patients with abnormal coagulation (PT International Normalized Ratio >1.2 or activated Partial Thromboplastin Time>45 sec)
9. Patients with uncontrolled diabetes
10. Treatment with aspirin or antithrombotic agents within 7days before operation
11. Treatment with anticoagulant drug
12. History of preoperative stress dose steroid treatment
13. Patients who the investigators believe will be ineligible for participation in the clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | within a month
Amount of drain at postoperative period | within a month

SECONDARY OUTCOMES:
Operation time | within 2 months
Transfusion | within 2 months
Inflammatory factors (Serum C-Reactive Protein and cytokines, ascites cytokines) | within 2 months
Postoperative hospital stay | within 2 months
4. Postoperative hospital stay Complications | within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Han-Kwang Yang, M.D., Ph.D., Principal Investigator — Seoul National University Hospital, Seoul, Korea, Republic of.
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Oh SY, Choi B, Lee KG, Choe HN, Lee HJ, Suh YS, Kong SH, Lee HJ, Kim WH, Yang HK. Ultrasonically Activated Shears Reduce Blood Loss without Increasing Inflammatory Reactions in Open Distal Gastrectomy for Cancer: A Randomized Controlled Study. Ann Surg Oncol. 2017 Feb;24(2):494-501. doi: 10.1245/s10434-016-5518-3. Epub 2016 Sep 9. PMID 27613551